CLINICAL TRIAL: NCT00038714
Title: A Phase II Trial of SGN-00101 In The Treatment of Pediatric Recurrent Respiratory Papillomatosis
Brief Title: A Trial Study of SGN-00101 in Treating Pediatric Patients With Recurrent Respiratory Papillomatosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nventa Biopharmaceuticals Corporation (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Stressgen SGN-00101-0005; SGN-00101-0005
Record Dates: First submitted 2002-06-04; First posted 2002-06-05 (Estimated); Last update posted 2007-06-27 (Estimated); Status verified 2007-06

CONDITIONS: Papilloma; Recurrent Respiratory Papillomatosis
Keywords: HPV; Papilloma
MeSH Terms: conditions — Papilloma; Recurrent respiratory papillomatosis

INTERVENTIONS:
Drug: SGN-00101

SUMMARY:
Recurrent Respiratory Papillomatosis (RRP) causes wart-like lesions along the throat area and can obstruct the airway or become malignant. The cause has been related to specific types of Human Papillomavirus (HPV). The purpose of the study is to assess the clinical effectiveness of a trial drug, SGN-00101, in children with RRP and also assess its safety.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 2 and 18 yrs old, inclusive, who has documented RRP.
* Patients with documented RRP
* Subject is surgically debulked within 7 days before the first dose of SGN-00101.
* Subject has had at least 4 debulking surgeries for RRP, had no intersurgical intervals greater than 84 days during the period of the last 4 surgeries.
* Subject is free of life threatening or serious concomitant disorders other than the disease under study.
* Females of childbearing potential must have a negative pregnancy test and must be practicing an effective/appropriate method of birth control as determined by the Investigator.

Exclusion Criteria:

* Subject has disease or status that causes compromise of the immune system.
* Subject has a history of ionizing radiation therapy to the respiratory tract.
* Patient has used concomitant medications that may suppress the immune system.
* Subject has received any specific or non-specific immunotherapy intended as treatment for their RRP (i.e. mumps vaccine injected intralesionally) within 9 months prior to Week 0 of this study.
* Subject has participated in a past study with SGN-00101
* Pregnancy and lactation.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 27 (Estimated)
Dates: Start 2001-11; Study Completion 2004-01

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - University of Arkansas for Medical Sciences, Arkansas Children's Hospital, Little Rock, Arkansas
  - Nemour's Childrens Clinic, Division of Pediatric Oncology, Jacksonville, Florida
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Fairview University Medical Center, University of Minnesota, Minneapolis, Minnesota
  - University Hospitals of Cleveland, Cleveland, Ohio
  - University of Texas, Southwestern Medical School, Dallas, Texas
  - Children's Hospital of the King's Daughters, Norfolk, Virginia